CLINICAL TRIAL: NCT05265273
Title: An Open-Label Uncontrolled Multicenter Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Activity of Nipocalimab in Children Aged 2 to Less Than 18 Years With Generalized Myasthenia Gravis
Brief Title: A Study of Nipocalimab in Children Aged 2 to Less Than 18 Years With Generalized Myasthenia Gravis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109137; 80202135MYG2001 (Other: Janssen Research & Development, LLC); 2021-002479-20 (EudraCT Number); 2022-502539-21-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05221619 (Temporarily not available)
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Myasthenia Gravis
Keywords: Pediatric
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nipocalimab (Experimental): Participants age 2 to less than (<) 18 years of age (globally) and 8 to <18 years of age (for US sites only) will be divided into 2 cohorts as per their age-adolescents 12 to <18 years and children 2 to <12 years and will receive nipocalimab once every two weeks for 24 weeks. After Week 24, all participants will have the option to enroll in long term extension (LTE).
  Interventions: Drug: Nipocalimab

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered as an IV infusion.
  Other Names: M281/JNJ-80202135

SUMMARY:
The purpose of this study is to determine the effect of nipocalimab on total serum immunoglobulin G (IgG) in pediatric participants 2 to less than (<) 18 years of age (globally) and 8 to <18 years of age (for Unites Stated (US) sites only), the safety and tolerability of treatment with nipocalimab in children and adolescents and to evaluate the pharmacokinetics (PK) of nipocalimab in children and adolescents with generalized myasthenia gravis (gMG) who have an insufficient clinical response to ongoing, stable standard-of-care therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Age: For US sites only: 8 to < 18 years
* Diagnosis of myasthenia gravis (MG) with generalized muscle weakness meeting the clinical criteria for generalized myasthenia gravis (gMG) as defined by the Myasthenia Gravis Foundation of America (MGFA) Clinical Classification Class IIa/b, IIIa/b, or IVa/b at screening
* Has a positive serologic test for acetylcholine receptor (anti-AChR) antibodies or muscle-specific tyrosine kinase (anti-MuSK) antibodies at screening
* A participant using herbal, naturopathic, traditional Chinese remedies, ayurvedic or nutritional supplements, or medical marijuana (with a doctor's prescription) is eligible if the use of these medications is acceptable to the Investigator. These remedies must remain at a stable dose and regimen throughout the study
* Has sufficient venous access to allow drug administration by infusion and blood sampling as per the protocol
* Participants should have a body weight and body mass index between 5th and 95th percentile for age and sex. Obese participants greater than 95th percentile and underweight participants below 5th percentile may participate following medical clearance
* A female of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at Screening and a negative urine pregnancy test at Day 1 prior to administration of study intervention

Key Exclusion Criteria:

* Has a history of severe and/or uncontrolled hepatic (example, viral/alcoholic/ autoimmune hepatitis/ cirrhosis/ and/or metabolic liver disease), gastrointestinal, renal, pulmonary, cardiovascular (including congenital heart diseases), psychiatric, neurological musculoskeletal disorder, any other medical disorder(s) (example, diabetes mellitus), risk factors for thrombosis events (example, a history of venous thromboembolism [VTE] or antiphospholipid syndrome, or a personal or family history of heritable coagulation disorder such as factor V leiden, protein S or protein C deficiency, atrial fibrillation/flutter, major orthopedic surgery or significant trauma that may increase the risk of VTE, is expected to be immobilized for prolonged periods of time), or has clinically significant abnormalities in screening laboratory, that might interfere with participant's full participation in the study, and/ or might jeopardize the safety of the participant or the validity of the study results
* Has any confirmed or suspected clinical immunodeficiency syndrome not related to treatment of his/her generalized myasthenia gravis (gMG), or has a family history of congenital or hereditary immunodeficiency unless confirmed absent in the participant
* Has had a thymectomy within 12 months prior to screening, or thymectomy is planned during the Active treatment Phase of the study
* Has shown a previous severe immediate hypersensitivity reaction, such as anaphylaxis to therapeutic proteins (example, monoclonal antibodies)
* Has experienced myocardial infarction, unstable ischemic heart disease, or stroke within 12 weeks of screening

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Total Serum Immunoglobulin-G (IgG) Levels | Up to 3 years
  Change from baseline in total serum IgG levels were reported.
Number of Participants with Infectious Adverse Events (AEs) | Up to 3 years
  Number of participants with infectious AEs will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Serious AEs (SAEs) | Up to 3 years
  Number of participants with SAEs will be reported. A SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect, is suspected transmission of any infectious agent via a medicinal product, is medically important to prevent one of the outcomes listed above.
Number of Participants with Adverse Events of Special Interests (AESIs) | Up to 3 years
  Number of participants with AESIs will be reported. Treatment-emergent AEs associated with the following situations are considered an AESI: a) infections that are severe or require intravenous (IV) anti-infective or operative/invasive intervention; b) hypoalbuminemia with albumin less than (<)20 grams per liter (g/L) [<] 2.0 grams per deciliter [g/dL]) c) opportunistic infections and d) Serious and non-serious deep-vein thrombosis (DVT) and/or pulmonary embolism (PE). Any AE occurring at or after the initial administration of study intervention through end of study is treatment emergent.
Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to 3 years
  Number of participants with abnormalities in clinical laboratory tests (including chemistry, hematology, coagulation, and urinalysis) will be reported.
Number of Participants with Abnormalities in Vital Signs | Up to 3 years
  Number of participants with abnormalities in vital signs including sitting pulse/heart rate, sitting systolic and diastolic blood pressure, and oral temperature (degrees Celsius) will be reported.
Number of Participants with Abnormalities in Physical Examination | Up to 3 years
  Number of participants with abnormalities in physical examinations including height, weight, assessments of the skin, head, eyes, ears, nose, throat, neck, thyroid, lungs, heart, abdomen, lymph nodes and extremities will be reported.
Serum Concentration of Nipocalimab over Time | Up to 3 years
  Serum samples will be analyzed to determine concentrations of nipocalimab using a validated, specific, and sensitive immunoassay method.
Clearance (CL) of Nipocalimab | Up to 3 years
  CL is defined as the volume of serum from which nipocalimab is completely removed per unit time.
Volume of Distribution (V) of Nipocalimab | Up to 3 years
  V is defined as the representation of nipocalimab's propensity to either remain in the serum or redistribute to other tissue compartments.
Half-life (t1/2) of Nipocalimab | Up to 3 years
  t1/2 is defined as the time it takes for nipocalimab's active substance in the body to reduce by half.
Steady-state Peak Concentration (Cpeak,ss) of Nipocalimab | Up to 3 years
  Cpeak,ss is defined as the peak serum concentration of nipocalimab at steady state.
Steady-state Trough concentration (Ctrough,ss) of Nipocalimab | Up to 3 years
  Ctrough,ss will be reported. It is defined as the observed serum concentration of nipocalimab just prior to the beginning of a dosing interval at steady state.
Steady-state Area Under the Curve (AUCss) of Nipocalimab | Up to 3 years
  AUCss is defined as the area under the curve for nipocalimab at steady state.

SECONDARY OUTCOMES:
Change from Baseline in Myasthenia Gravis -Activities of Daily Living (MG-ADL) Score | Up to 3 years
  Change from baseline in MG-ADL score will be reported. The MG-ADL score provides a rapid assessment of the participant's myasthenia gravis (MG) symptom severity. Eight functions (talking, chewing, swallowing, breathing, impairment of ability to brush teeth or comb hair, impairment of ability to arise from a chair, double vision, eyelid droop) are rated on a 4-point scale: 0 (no impairment) to 3 (severe impairment). The total score will be sum of eight function scores and can range from 0 to 24. A higher score indicates greater symptom severity.
Change in the Quantitative Myasthenia Gravis (QMG) Score | Up to 3 years
  The QMG score is a standardized quantitative strength assessment comprising 13 components (and is administered by a trained qualified healthcare professional [HCP] eg, physician, physician assistant, nurse practitioner, nurse). The quantitative results of each strength component are mapped to the following 4-point scale: 0 equals to (=) none, 1 = mild, 2 = moderate and 3 = severe. The total score will be sum of 13 components scores and can range from 0 to 39. A higher score indicates greater weakness.
European Quality of Life 5-Dimension Youth (EQ-5D-Y) Tool Score | Up to 3 years
  The EQ-5D-Y is a standardized child friendly instrument for use as a measure of health status, primarily designed for self-completion by children and adolescents, or via a proxy version to be completed by the child's caregiver. The EQ-5D-Y descriptive system comprises the following 5 dimensions: Mobility, looking after myself (washing and dressing), usual activities, pain or discomfort and feeling worried or unhappy. Each of the 5 dimensions is divided into 3 levels of perceived problems (Level 1 indicating no problem, Level 2 indicating some problems, Level 3 a lot of problems).
Neurological Quality of Life (Neuro-QoL) Pediatric Fatigue Score | Up to 3 years
  The Neuro-QoL pediatric fatigue score will be used to assess the impact of fatigue in participants aged 10 to less than (<) 18 years. The participant will rate each of the 11 items on a 5-point scale. Higher scores indicate greater fatigue.
Patient Global Impression of Severity (PGI-S) Score | Up to 3 years
  The PGI-S score will be used to assess the severity of fatigue due to generalized myasthenia gravis (gMG) in participants aged 10 to < 18 years. Participants will be asked to rate their fatigue over the past 7 days using the following 5-point scale: 1 = None, 2 = Mild, 3 = Moderate, 4 = Severe, and 5 = Very severe. Higher scores indicate greater severity of fatigue.
Patient Global Impression of Change (PGI-C) Score | Up to 3 years
  The PGI-C score will be used to assess if there has been an improvement or decline in patient-reported fatigue since the beginning of the treatment in participants aged 10 to <18 years. Participants will be asked to rate their current fatigue as compared to when they started the study, using the following 7-point scale: 1 = Much better, 2 = Moderately better, 3 = A little better, 4 = No change, 5 = A little worse, 6 = Moderately worse, and 7 = Much worse. Higher scores indicate greater change in overall fatigue.
Number of Participants with Anti-Drug Antibodies [ADAs] to Nipocalimab | Up to 3 years
  Number of participants with ADAs to nipocalimab will be reported.
Number of Participants with Neutralizing Antibodies (NAbs) to Nipocalimab | Up to 3 years
  Number of participants with NAbs to nipocalimab will be reported.
Number of Participants with Vaccine Antibody Titers to Diphtheria or Tetanus | Up to 3 years
  Number of participants with vaccine antibody titers to diphtheria or tetanus will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (19):
- United States (11):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of South Florida Morsani Center for Advanced Healthcare, Tampa, Florida
  - University of Kansas Medical Center, Lawrence, Kansas
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Penn State Milton S Hershey Medical Ctr, Hershey, Pennsylvania
  - Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Japan (6):
  - Nagano Children's Hospital, Azumino-shi
  - Chiba University Hospital, Chiba
  - University of Miyazaki Hospital, Miyazaki
  - Hyogo College of Medicine Hospital, Nishinomiya-Shi
  - Saitama Prefecture Children's Medical Center, Saitama Shi
  - Tokyo Women's Medical University Hospital, Shinjuku-ku
- Leiden University Medical Center, Leiden, Netherlands
- Uniwersyteckie Centrum Kliniczne, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency